CLINICAL TRIAL: NCT03901131
Title: PROMES: PROspective, Non-Interventional, Observational, Longitudinal Study to Describe the Safety Profile of MESIGYNA® (Norethisterone Enantate 50 mg and Estradiol Valerate 5 mg) as a Contraceptive Method for Women in Reproductive Age at the Outpatient Clinic
Brief Title: PROMES: A Clinical Study in Which Researchers Want to Learn More About the Safety Profile of MESIGYNA (Norethisterone Enantate 50 mg and Estradiol Valerate 5 mg) Used as a Medication to Prevent Pregnancy for Adult Women in Reproductive Age in the Peruvian Population at the Outpatient Clinic.
Acronym: PROMES
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19243
Record Dates: First submitted 2019-02-20; First posted 2019-04-03 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Contraceptive
MeSH Terms: interventions — norethindrone enanthate; Estradiol; estradiol, norethindrone drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAY98-7040: Female adult patients of reproductive age, who want to use a contraceptive method, will be enrolled after the investigator has made the decision for treatment with Mesigyna.
  Investigators should prescribe Mesigyna for medically approved indications as per the label of the medicine locally approved.
  Interventions: Drug: Norethisterone enantate/estradiol valerate (Mesigyna, BAY98-7040)

INTERVENTIONS:
Drug: Norethisterone enantate/estradiol valerate (Mesigyna, BAY98-7040) — Follow clinical administration

SUMMARY:
Clinical study in which researchers want to learn more about the safety profile of MESIGYNA used as a medication in routine clinical practice to prevent pregnancy. In order to find this out researchers will collect historic and treatment related data during initial visit and follow-up visits of adult women in reproductive age in the Peruvian population at the outpatient clinic. Mesigyna is a combined injectable birth control medication (norethindrone ethanate (50 mg) and estradiol valerate (5 mg)) for women given monthly.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients,18 to 45 years old with a Mesigyna prescription
* Women for whom the decision to initiate contraception with Mesigyna was made as per investigator's routine practice
* Signed Informed Consent

Exclusion Criteria:

* Women participating in an investigational program with interventions outside of routine clinical practice
* Hypersensitivity to norethisterone enantate or estradiol valerate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who have been prescribed Mesigyna in Peru.
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events and Serious Adverse Events | Up to 6 months

SECONDARY OUTCOMES:
The number of injections | Up to 6 months
Number of injections | Up to 6 months
Frequency of injections | Up to 6 months
Comorbidities associated to greater incidence of AE and SAE | Up to 6 months
  The associated factors for AE for contraceptives are headaches, acne, obesity, hypertension, breast tenderness, dysmenorrhea, nausea. This could get worse with the use of contraceptives.

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Peru

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/